CLINICAL TRIAL: NCT03944239
Title: Safety and Efficacy of Subretinal Transplantation of Clinical Human Embryonic Stem Cell Derived Retinal Pigment Epitheliums in Treatment of Retinitis Pigmentosa
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qi Zhou (Other Government)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor-Investigator, Qi Zhou, Director of Institute of zoology, chinese academy of sciences, and vice president of medical school， University of chinese academy of sciences, Chinese Academy of Sciences
Organization: Chinese Academy of Sciences (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ChineseASZQ-002
Record Dates: First submitted 2018-12-27; First posted 2019-05-09 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- retinal pigment epitheliums transplantation (Experimental): Transplant clinical-grade hESC derived retinal pigment epitheliums into subretinal of patients with retinitis pigmentosa.The dosage is 150000.
  Interventions: Biological: Retinal pigment epitheliums transplantation

INTERVENTIONS:
Biological: Retinal pigment epitheliums transplantation — Subretinal transplantation of clinical human embryonic stem cell derived retinal pigment epitheliums.

SUMMARY:
This project intends to transplant a clinical level human embryonic stem cells derived retinal pigment epithelium into subretinal space to treat eetinitis pigmentosa(RP) diseases. Through the statistical analysis EDTRS, BCVA, OCT, ERG, Fluorescein angiography, Ophthalmic AB ultrasound changes between before and after the treatment to assess the efficacy and safety 0f RPE transplants to treat RP disease.

DETAILED DESCRIPTION:
This project intends to transplant a clinical level human embryonic stem cells derived retinal pigment epithelium into subretinal space to treat eetinitis pigmentosa(RP) diseases. Through the statistical analysis EDTRS, BCVA, OCT, ERG, Fluorescein angiography, Ophthalmic AB ultrasound changes between before and after the treatment to assess the efficacy and safety 0f RPE transplants to treat RP disease.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and under 80 years of age, both gender, in good health.
* Clinical diagnosis of retinitis pigmentosa, the results of eye electrophysiological examination accord with retinitis pigmentosa.
* The BCVA of target eye will not be better than 20/400.
* The BCVA of contralateral eye is not worse than 20/400.
* Diopter is smaller than 8.00 D, axial 28 mm or less.
* Voluntary as test subjects, signed informed consent, regular follow-up will be effected according to the specified time.

Exclusion Criteria:

* Subject with other additional retinal diseases, like diabetic or hypertensive retinopathy vascular diseases.
* Target eye ever have had a eye surgery;
* Subject with active serious diseases of the digestive system, liver kidney impairment (ALT/AST) > 1.5 or any known liver disease, creatine > 1.3 mg/dL) and/serious temic diseases, such as cardiovascular tem, respiratory tem, nervous tem, endocrine tem urogenital tem diseases, etc.), the history of malignancy;
* Have been ready for pregnancy during test, are lactating women;
* Ready to birth of men during the test;
* Subject with any immunodeficiency;
* Subject in the immunosuppressive therapy in the current;
* Subject with the tacrolimus or other large ring lactone class drug allergies;
* Participate in any clinical subjects in nearly six months;
* Has a history of alcohol or illicit drug abuse;
* Poor adherence to complete studies;
* Researchers believe that there may be an increased risk subjects or interfere with the clinical trials of any situation (such as when a patient is prone to mental tension, depression, mental illness, cognitive dysfunction, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events occurred within 1 year after transplantation | one year
  The occurrence of adverse events (AE), severe adverse events (SAE), treatment-related adverse events (TEAE), and clinically significant vital signs during the study period.

SECONDARY OUTCOMES:
Improvement of visual function | one year
  The changes of BCVA and EDTRS were observed one year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Qi, Doctor, Principal Investigator — Institute of Zoology, Chinese Academy of Sciences
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University, Beijing, Beijing Municipality, China